CLINICAL TRIAL: NCT02439983
Title: A Randomized, Double-blind, Placebo-controlled Study Investigating the Effects of a Proprietary Nutritional Supplement on Brain Health
Brief Title: Brain Imaging Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 14-PHX-0002
Record Dates: First submitted 2015-04-30; First posted 2015-05-12 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Brain Health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Proprietary Nutritional Supplement (Experimental)
  Interventions: Dietary Supplement: Proprietary Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: Proprietary Nutritional Supplement — 2 capsules taken by mouth with morning and evening meals.
  Arms: Proprietary Nutritional Supplement
Dietary Supplement: Placebo — 2 capsules taken by mouth with morning and evening meals.
  Arms: Placebo

SUMMARY:
The study is designed to evaluate the effects of the proprietary nutritional supplement on cognition, mood, and brain imaging parameters following a relatively short period of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female subjects will be included.
* Age between 40-60 years inclusive.
* Healthy subjects who, in the opinion of the investigator, are free of any medical conditions that might affect study measures.
* Eats 1 or fewer servings of fatty fish per week.
* BMI < 35

Exclusion Criteria:

* Current or past neurological illness.
* Substance abuse or dependence within the prior 60 days.
* Current depression (HAMD greater than 20) or anxiety disorder (HAMA greater than 18).
* Current or past history of psychiatric disorder.
* History of head trauma with loss of consciousness.
* Contraindication to brain MRI examination.
* Supplementation with Omega 3, fish oil, or other over the counter supplements including the other bioactive ingredients in the proprietary nutritional supplement, antioxidants and multi-vitamin mineral supplements for the previous 3 months.
* Plasma Omega3 Index >5% at screening visit.
* Subject has a known allergy or intolerance to any of the ingredients contained in the proprietary nutritional supplement or placebo.
* Subject is currently pregnant, planning to become pregnant, or is breastfeeding.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in MRI Brain scan | Change from Baseline MRI Brain scan at Day 42
  Determine differences in brain metabolism, brain connectivity, or brain structure. Highlight regional brain changes between pre and post chronic supplementation with a proprietary nutritional formula.

SECONDARY OUTCOMES:
Change in anxiety as measured by the Hamilton Anxiety Scale (HAM-A) | Change from Baseline anxiety at Day 42
Change in depression as measured by the Hamilton Depression Rating Scale (HAM-D) | Change from Baseline depression at Day 42
Change in mood as measured by the Profile of Mood States (POMS) | Change from Baseline mood at Day 42
Change in memory as measured by Logical Memory I and II (subtests from the Wechsler Memory Scale- IV) | Change from Baseline memory at Day 42
Change in fluency as measure by Letter and Category Fluency test | Change from Baseline fluency at Day 42
Change in Chemistry panel | Change from Baseline Chemistry panel at Day 42
Change in RBC fatty acid profile | Change from Baseline RBC fatty acid profile at Day 42
Change in Gene expression | Change from Baseline Gene expression at Day 42
Measurement of polyphenol metabolites in saliva | Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Yurgelun-Todd, Ph.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah - Brain Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Mastaloudis A, Sheth C, Hester SN, Wood SM, Prescot A, McGlade E, Renshaw PF, Yurgelun-Todd DA. Supplementation with a putative calorie restriction mimetic micronutrient blend increases glutathione concentrations and improves neuroenergetics in brain of healthy middle-aged men and women. Free Radic Biol Med. 2020 Jun;153:112-121. doi: 10.1016/j.freeradbiomed.2020.04.017. Epub 2020 Apr 23. PMID 32335159